CLINICAL TRIAL: NCT01570933
Title: Feasibility Study Over the Neurally Adjusted Ventilatory Assist (NAVA) Mode in Noninvasive Ventilation After Cardiac Surgery in Infants.
Brief Title: Feasibility Study Over the NAVA Mode in Noninvasive Ventilation After Cardiac Surgery in Infants.
Acronym: NIVNAVA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SIP2011
Record Dates: First submitted 2012-03-06; First posted 2012-04-04 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Heart Defects, Congenital; Surgery
Keywords: cardio-pulmonary bypass
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Interactive Ventilatory Support; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NAVAfirst (Experimental): Starting crossover by NIVnava mode
  Interventions: Device: NivNava
- Cpap first (Active Comparator): Start crossover by Cpap on nasal canula
  Interventions: Device: Cpap

INTERVENTIONS:
Device: NivNava — Non-invasive Nava ventilation mode on nasal cannula
  Other Names: Neurally adjusted ventilatory assist
  Arms: NAVAfirst
Device: Cpap — nasal Cpap on nasal cannula
  Other Names: InfantFlow(R), CareFusion(R), SanDiego, Ca, USA
  Arms: Cpap first

SUMMARY:
Neonates who underwent cardiac surgery with cardiopulmonary bypass almost always require non-invasive respiratory support (NIV) in relay to conventional ventilation. Current nasal interfaces do not generally allow synchronised bilevel ventilation. NIV-NAVA mode allows, through an oesophageal catheter, to record the electrical activity of the diaphragm and thereby synchronize breaths from the ventilator on the inspiratory efforts of the child. Moreover, the pressure support delivered by the ventilator may be proportional to the diaphragmatic effort developed by the child. This mode, associated with the interface Miniflow®, could increase the comfort of the child by allowing a more efficient synchronization and reducing its respiratory work. To our knowledge, this ventilation mode with this interface has not been evaluated in the postoperative period of cardiac surgery in the newborns. The purpose of this study is to evaluate the feasibility of this ventilatory mode and evaluate its influence on ventilatory parameters of this category of infants.

DETAILED DESCRIPTION:
Study Design:

Single centre prospective crossover study

Study Objectives:

Main objectives:

* Assessment of the feasibility of non invasive ventilation in NIV-NAVA mode via Miniflow® interface in infants of less than 3.5 kg after cardiac surgery with cardiopulmonary bypass.
* Evaluation of the following parameters:

  * Implementation of the interface
  * Air leaks
  * Placement and contention of oesophageal probe
  * Quality of synchronization
  * Obstruction of the probe
  * Risk of nasal wounds

Secondary objectives:

* Comparison of ventilation parameters between nasal Continuous Positive Airway Pressure (nCPAP) mode and NIV-NAVA mode
* Evaluation of the following parameters:

  * Breathing rhythm
  * Tidal volume
  * PEEP
  * Inspiratory pressure
  * FiO2
  * PaO2
  * PaCO2
  * pH
* Evolution of EAdi min and EAdi max parameters in NIV-NAVA mode (EAdi : diaphragmatic electric activity)

Conduct of the study:

First phase: placement of EADI catheter and extubation

When extubation criteria are met, the oesophageal EADI catheter is placed according to the manufacturer's instructions. The ventilation mode is then switched to Pressure Support Mode with the same Peep as in the previous mode and a pressure support of 10 cmH2O.

During 30 minutes, trends in respiratory rate, tidal volume, PEEP, inspiratory pressure, FiO2, EADI min, EADi max are recorded.

After 30 minutes, an arterial blood gas analysis is performed to determine the values of PaCO2, PaO2 and pH before randomization.

The child is extubated according to the procedures of the service and the non-invasive ventilation relay is introduced through the Miniflow® interface with nasal prongs adapted to the morphology of the child. An adrenaline nebulisation can be given before starting NIV in case of respiratory distress due to laryngeal oedema.

Second phase: nCPAP or NIV-NAVA

Following randomisation, the child is included in the "nCPAP first" arm or "NIV-NAVA first" arm and is ventilated in the designated mode for 30 minutes. During the first 15 minutes, the ventilation parameters are adapted according to the procedures below:

nCPAP parameters adaptation:

* PEEP and FiO2 as previously set in invasive ventilation;
* FiO2 according to target SpO2 values of the child and/or 10% higher than FiO2 in invasive ventilation mode;
* PEEP between 4-6 cmH2O in order to minimize respiratory efforts.

NIV-NAVA parameters adaptation:

* PEEP and FiO2 as previously set in invasive ventilation;
* Adaptation of the NIV-NAVA level to reach a EADi level equal to the mean EADi level over the last 5 minutes of the invasive mode. Inspiratory pressure and tidal volume are limited respectively to 30 cmH2O and 8 ml/kg.
* FiO2 according to target SpO2 values of the child and/or 10% higher than FiO2 in invasive ventilation mode ;
* PEEP between 4-6 cmH2O in order to minimize respiratory efforts.

Over the last 15 minutes of this ventilation mode, trends in respiratory rate, tidal volume, PEEP, inspiratory pressure, FiO2, EADI min, EADi max are recorded.

On Minutes M16, M21 and M29 in NIV-NAVA mode, synchronisation data are recorded : auto-triggering, double triggering, inspiration beginning and ending.

After 30 minutes, an arterial blood gas analysis is performed to determine the evolution of the values of PaCO2, PaO2 and pH.

At any time, if the re-intubation criteria are met, the child is re-intubated and returned to conventional ventilation. He is then excluded of the study.

Third phase: nCPAP or NIV-NAVA

The ventilation mode is changed from nCPAP to NIV-NAVA or from NIV-NAVA to nCPAP. The adaptation protocol and the recorded parameters are the same as in the second phase.

After 30 minutes, an arterial blood gas analysis is performed to determine the evolution of the values of PaCO2, PaO2 and pH.

At any time, if the re-intubation criteria are met, the child is re-intubated and returned to conventional ventilation. He is then excluded of the study.

Fourth phase: end of the study

The study concludes at the end of the third phase. The child is left in the better tolerated ventilation mode, as judged by the clinician.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≤ 5 kg
* Postoperative period of cardiac surgery with cardiopulmonary bypass (max 10 days after surgery)
* Conventional ventilation
* Agreement with the extubation criteria
* Arterial line

Exclusion Criteria:

* High frequency oscillation ventilation
* Extubation criteria not fulfilled
* Proven or suspected sepsis
* Absence of arterial line
* Oesophageal pathology (Excepted gastro-oesophageal reflux)

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the percentage of asynchronies during the nava mode | from minute zero to minute 90
  One of the aims of the NAVA mode is to provide better synchronization between the child's breathing needs and the breathing cycles given by the ventilator. By comparing the EDI curve (electric activity of the diaphragm of the child) and the flow and pressure curves of the ventilator, it is possible to determine the percentage of asynchronies during the nava mode

SECONDARY OUTCOMES:
Comparison of breathing rhythm between nasal Continuous Positive Airway Pressure (nCPAP) mode and NIV-NAVA mode | from minute zero to minute 90
Comparison of PEEP (positive end expiratory pressure) between nasal Continuous Positive Airway Pressure (nCPAP) mode and NIV-NAVA mode | from minute zero to minute 90
Comparison of Inspiratory Pressure between nasal Continuous Positive Airway Pressure (nCPAP) mode and NIV-NAVA mode | from minute zero to minute 90
Comparison of FiO2 between nasal Continuous Positive Airway Pressure (nCPAP) mode and NIV-NAVA mode | from minute zero to minute 90
Comparison of PaO2 between nasal Continuous Positive Airway Pressure (nCPAP) mode and NIV-NAVA mode | from minute zero to minute 90
Comparison of PaCO2 between nasal Continuous Positive Airway Pressure (nCPAP) mode and NIV-NAVA mode | from minute zero to minute 90
Comparison of blood pH between nasal Continuous Positive Airway Pressure (nCPAP) mode and NIV-NAVA mode | from minute zero to minute 90

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Houtekie, md, Principal Investigator — Cliniques Universitaires Saint-LUc, Brussels
Locations (1):
- Cliniques Univeristaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Houtekie L, Moerman D, Bourleau A, Reychler G, Detaille T, Derycke E, Clement de Clety S. Feasibility Study on Neurally Adjusted Ventilatory Assist in Noninvasive Ventilation After Cardiac Surgery in Infants. Respir Care. 2015 Jul;60(7):1007-14. doi: 10.4187/respcare.03624. Epub 2015 Feb 17. PMID 25691764